CLINICAL TRIAL: NCT00003816
Title: Allogeneic Blood or Marrow Transplantation for Hematologic Malignancy and Aplastic Anemia
Brief Title: Combination Chemotherapy and Donor Stem Cell Transplant in Treating Patients With Aplastic Anemia or Hematologic Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP 98-15; RP 98-15 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Nonmalignant Neoplasm; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent cutaneous T-cell non-Hodgkin lymphoma; Burkitt lymphoma; Waldenstrom macroglobulinemia; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; polycythemia vera; essential thrombocythemia; refractory anemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; intraocular lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; primary myelofibrosis; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes; aplastic anemia; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Thrombocythemia, Essential; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Intraocular Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Primary Myelofibrosis; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities; Anemia, Aplastic | interventions — Antilymphocyte Serum; Busulfan; Carboplatin; Cyclophosphamide; Etoposide; fludarabine phosphate; Melphalan; Thiotepa; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Regimen 1 (Experimental): Patients receive busulfan IV over 2 hours every 6 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2.
  Interventions: Drug: busulfan; Drug: cyclophosphamide
- Regimen 2 (Experimental): Patients receive cyclophosphamide IV over 2 hours on days -5 to -2 and anti-thymocyte globulin IV over 4-8 hours on days -5 to -3.
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide
- Regimen 3 (Experimental): Patients receive cyclophosphamide IV over 2 hours on days -5 and -4 and total-body irradiation (TBI) twice daily on days -3 to -1.
  Interventions: Drug: cyclophosphamide; Radiation: total-body irradiation
- Regimen 4 (Experimental): Patients receive fludarabine IV over 30 minutes on days -6 to -2 and melphalan IV over 1 hour on days -3 and -2.
  Interventions: Drug: fludarabine phosphate; Drug: melphalan
- Regimen 5 (Experimental): Patients receive etoposide IV over 26 hours beginning on day -5, cyclophosphamide IV over 2 hours on day -4, and TBI twice daily on days -3 to -1.
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Radiation: total-body irradiation
- Regimen 6 (Experimental): Patients receive cyclophosphamide IV over 24 hours, carboplatin IV over 24 hours, and thiotepa IV over 24 hours on days -7 to -4.
  Interventions: Drug: carboplatin; Drug: cyclophosphamide; Drug: thiotepa
- Regimen 7 (Experimental): Patients receive fludarabine IV over 30 minutes on days -5 to -1 and anti-thymocyte globulin IV over 4-8 hours on days -5 to -2.
  Interventions: Biological: anti-thymocyte globulin; Drug: fludarabine phosphate
- Regimen 8 (Experimental): Patients receive cyclophosphamide IV over 2 hours on days -5 and -4, TBI twice daily on days -3 to -1, and anti-thymocyte globulin IV over 4-8 hours on days -3 to -1.
  Interventions: Biological: anti-thymocyte globulin; Drug: cyclophosphamide; Radiation: total-body irradiation
- Regimen 9 (Experimental): Patients receive busulfan IV over 2 hours every 6 hours and anti-thymocyte globulin IV over 4-8 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2.
  Interventions: Biological: anti-thymocyte globulin; Drug: busulfan; Drug: cyclophosphamide

INTERVENTIONS:
Biological: anti-thymocyte globulin — Given IV
  Arms: Regimen 2; Regimen 7; Regimen 8; Regimen 9
Drug: busulfan — Given IV
  Arms: Regimen 1; Regimen 9
Drug: carboplatin — Given IV
  Arms: Regimen 6
Drug: cyclophosphamide — Given IV
  Arms: Regimen 1; Regimen 2; Regimen 3; Regimen 5; Regimen 6; Regimen 8; Regimen 9
Drug: etoposide — Given IV
  Arms: Regimen 5
Drug: fludarabine phosphate — Given IV
  Arms: Regimen 4; Regimen 7
Drug: melphalan — Given IV
  Arms: Regimen 4
Drug: thiotepa — Given IV
  Arms: Regimen 6
Radiation: total-body irradiation — Given twice daily for 3 days
  Arms: Regimen 3; Regimen 5; Regimen 8

SUMMARY:
RATIONALE: Giving chemotherapy drugs and total-body irradiation before a donor stem cell helps stop the growth of cancer or abnormal cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. It is not yet known which combination chemotherapy regimen is most effective when given before a donor stem cell transplant in treating aplastic anemia or hematologic cancer.

PURPOSE: This phase II/III trial is studying different combination chemotherapy regimens to compare how well they work when given before donor stem cell transplant in treating patients with aplastic anemia or hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the morbidity, mortality, and overall outcome of patients with severe aplastic anemia or hematologic malignancy treated with standard vs novel conditioning regimens followed by allogeneic stem cell transplantation.
* Examine the influence of donor histocompatibility on outcome by comparing matched/related, mismatched/related (with or without T-cell depletion), and matched/unrelated transplants with stratification for type of preparative regimen.
* Ensure that patients with uncommon diagnoses will be treated in a uniform fashion with the best therapy available.

OUTLINE: Patients are stratified according to risk of relapse (standard-risk: acute leukemia in first complete remission, chronic myelogenous leukemia in first chronic phase, lymphoma in sensitive first relapse or second remission, primary or untreated myelodysplastic syndromes, or untreated severe aplastic anemia vs high-risk: all others).

Patients are assigned to one of the following conditioning regimens based on diagnosis, risk of relapse, and donor relatedness:

* Regimen 1: Patients receive busulfan IV over 2 hours every 6 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2.
* Regimen 2: Patients receive cyclophosphamide IV over 2 hours on days -5 to -2 and anti-thymocyte globulin IV over 4-8 hours on days -5 to -3.
* Regimen 3: Patients receive cyclophosphamide IV over 2 hours on days -5 and -4 and total-body irradiation (TBI) twice daily on days -3 to -1.
* Regimen 4: Patients receive fludarabine IV over 30 minutes on days -6 to -2 and melphalan IV over 1 hour on days -3 and -2.
* Regimen 5: Patients receive etoposide IV over 26 hours beginning on day -5, cyclophosphamide IV over 2 hours on day -4, and TBI twice daily on days -3 to -1.
* Regimen 6: Patients receive cyclophosphamide IV over 24 hours, carboplatin IV over 24 hours, and thiotepa IV over 24 hours on days -7 to -4.
* Regimen 7: Patients receive fludarabine IV over 30 minutes on days -5 to -1 and anti-thymocyte globulin IV over 4-8 hours on days -5 to -2.
* Regimen 8: Patients receive cyclophosphamide IV over 2 hours on days -5 and -4, TBI twice daily on days -3 to -1, and anti-thymocyte globulin IV over 4-8 hours on days -3 to -1.
* Regimen 9: Patients receive busulfan IV over 2 hours every 6 hours and anti-thymocyte globulin IV over 4-8 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2.

All patients then receive donor stem cell infusions on day 0. Some patients may undergo involved-field radiotherapy 4-8 weeks after transplant.

Patients will be taken off study after a minimum of 4 years of follow up.

PROJECTED ACCRUAL: At least 405 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Severe aplastic anemia as defined by either of the following:

    * Marrow cellularity (< 25% [or 25-50% cellularity with < 30% of remaining cells hematopoietic in origin])
    * At least 2 of the following abnormal peripheral blood counts:

      * Reticulocyte count < 1% (corrected for hematocrit)
      * Platelet count < 20,000/mm^3
      * Neutrophil count < 500/mm^3
  * Histologically confirmed hematologic malignancy, including any of the following:

    * Acute leukemia

      * Resistant or recurrent disease after combination chemotherapy with at least one standard regimen OR in first remission and at high risk of relapse
      * Acute myeloid leukemia (AML) (antecedent myelodysplastic syndromes [MDS], secondary AML, or high-risk cytogenetic abnormalities)
      * Acute lymphoblastic leukemia (ALL) (high-risk cytogenetic abnormalities)
    * Chronic myeloid leukemia (CML)

      * Chronic phase, accelerated phase, or blast phase
    * Myeloproliferative disorders or MDS, including any of the following:

      * Myelofibrosis
      * Polycythemia vera*
      * Essential thrombocythemia*
      * Refractory anemia
      * Refractory anemia with excess blasts
      * Refractory anemia with excess blasts in transformation
      * Chronic myelomonocytic leukemia NOTE: * Only if transformed to AML or MDS
    * Lymphoproliferative disease

      * Recurrent or persistent, symptomatic disease after first-line chemotherapy, including any of the following:

        * Chronic lymphocytic leukemia (CLL) (≥ 20% marrow involvement)
        * Waldenstrom macroglobulinemia
        * Low-grade non-Hodgkin lymphoma
    * Intermediate or high-grade non-Hodgkin lymphoma, meeting 1 of the following criteria:

      * Resistant or recurrent disease after combination chemotherapy with one standard regimen
      * Lymphoblastic lymphoma or small noncleaved cell lymphoma in first remission and at high risk of relapse
      * CNS disease
      * Bone marrow disease and LDH greater than 300
  * Solid tumor that would otherwise be treated on RPCI-DS-9115 (or equivalent autologous stem transplant protocol) AND has a syngeneic donor
* Autologous bone marrow transplant not possible (or desirable) due to 1 of the following:

  * History of marrow tumor
  * Inadequate marrow dose
  * Abnormal marrow histology or function prior to storage
  * Thrombocytopenia or leukopenia
  * Marrow cellularity < 20%
* Histocompatible donor identified

  * Well-matched donor, as defined by 1 of the following:

    * Family member matched for 5 or 6 HLA specificities (A, B, DR)*
    * Unrelated donor meeting compatibility criteria of the National Marrow Donor Program (matched for HLA A, B, and DRB1 antigens)*
    * Identical twin sibling
  * If a compatible cord blood donor is identified and there is no suitable unrelated donor available, patient may receive cord blood transplant NOTE: *Patients ≤ 25 years of age may be singly mismatched at the A or B loci

NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 4 to 70

Performance status:

* Zubrod 0-2 OR
* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin < 3 times normal (unless due to disease)
* Alkaline phosphatase < 3 times normal (unless due to disease)
* SGOT < 3 times normal (unless due to disease)
* Hepatitis B surface antigen negative
* No severe hepatic disease that would preclude study participation

Renal:

* Creatinine normal
* Creatinine clearance ≥ 50 mL/min
* No severe renal disease that would preclude study participation

Cardiovascular:

* Cardiac ventricular ejection fraction ≥ 50% by MUGA or echocardiogram
* No uncontrolled or severe cardiovascular disease (e.g., myocardial infarction, congestive heart failure, symptomatic angina, life threatening arrhythmia, or hypertension within the past 6 months)

Pulmonary:

* DLCO or DLVA ≥ 50% predicted (corrected for hemoglobin or alveolar ventilation)

Other:

* No serious concurrent medical or psychiatric illness
* No other serious organ dysfunction (unless due to underlying disease), including the following:

  * Uncontrolled bacterial, viral, or fungal infection
  * Uncontrolled peptic ulcer disease
  * Uncontrolled diabetes mellitus
* HIV negative
* Cytomegalovirus status known
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Pretransplant cytoreductive chemotherapy allowed for patients with relapsed or refractory disease

Endocrine therapy:

* Not specified

Radiotherapy:

* Not eligible for total-body irradiation if prior radiotherapy exceeded the following limits:

  * Mediastinum: 3,600 cGy
  * Heart: 3,600 cGy
  * Whole lungs: 1,200 cGy
  * Small bowel: 3,600 cGy
  * Kidneys: 1,200 cGy
  * Whole liver: 1,600 cGy
  * Cranial spinal: 3,600 cGy
  * Brain: 4,000 cGy
  * Retina: 4,000 cGy

Surgery:

* Not specified

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 1998-10-19 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L. McCarthy, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BuCy: Patients receive busulfan IV over 2 hours every 6 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2.
  busulfan: Given IV
  cyclophosphamide: Given IV
- CyTBI: Patients receive cyclophosphamide IV over 2 hours on days -5 and -4 and total-body irradiation (TBI) twice daily on days -3 to -1.
  cyclophosphamide: Given IV
  total-body irradiation: Given twice daily for 3 days
- FluMel: Patients receive fludarabine IV over 30 minutes on days -6 to -2 and melphalan IV over 1 hour on days -3 and -2.
  fludarabine phosphate: Given IV
  melphalan: Given IV
- VpCyTBI: Patients receive etoposide IV over 26 hours beginning on day -5, cyclophosphamide IV over 2 hours on day -4, and TBI twice daily on days -3 to -1.
  cyclophosphamide: Given IV
  etoposide: Given IV
  total-body irradiation: Given twice daily for 3 days
- Other: Patients receive cyclophosphamide IV over 2 hours on days -5 and -4, TBI twice daily on days -3 to -1, and anti-thymocyte globulin IV over 4-8 hours on days -3 to -1. OR Patients receive cyclophosphamide IV over 2 hours on days -5 to -2 and anti-thymocyte globulin IV over 4-8 hours on days -5 to -3. OR Patients receive cyclophosphamide IV over 24 hours, carboplatin IV over 24 hours, and thiotepa IV over 24 hours on days -7 to -4. OR Patients receive fludarabine IV over 30 minutes on days -5 to -1 and anti-thymocyte globulin IV over 4-8 hours on days -5 to -2. OR Patients receive busulfan IV over 2 hours every 6 hours and anti-thymocyte globulin IV over 4-8 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2.
Period: Overall Study
Arm/Group | BuCy | CyTBI | FluMel | VpCyTBI | Other
Started | 55 | 69 | 199 | 23 | 15
Completed | 55 | 69 | 199 | 23 | 15
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Other: Patients receive cyclophosphamide IV over 2 hours on days -5 to -2 and anti-thymocyte globulin IV over 4-8 hours on days -5 to -3. OR Patients receive cyclophosphamide IV over 24 hours, carboplatin IV over 24 hours, and thiotepa IV over 24 hours on days -7 to -4. OR Patients receive fludarabine IV over 30 minutes on days -5 to -1 and anti-thymocyte globulin IV over 4-8 hours on days -5 to -2. OR Patients receive cyclophosphamide IV over 2 hours on days -5 and -4, TBI twice daily on days -3 to -1, and anti-thymocyte globulin IV over 4-8 hours on days -3 to -1.
  OR Patients receive busulfan IV over 2 hours every 6 hours and anti-thymocyte globulin IV over 4-8 hours on days -7 to -4 and cyclophosphamide IV over 2 hours on days -3 and -2.
- Total: Total of all reporting groups
Arm/Group | BuCy | CyTBI | FluMel | VpCyTBI | Other | Total
Number analyzed (Participants) | 55 | 69 | 199 | 23 | 15 | 361
Age, Continuous [Median (Full Range); unit: years] | 46 [6 to 59] | 28 [4 to 50] | 48 [6 to 68] | 37 [8 to 55] | 41 [6 to 52] | 44 [4 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 80 | 7 | 4 | 139
  Male | 31 | 45 | 119 | 16 | 11 | 222
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 53 | 68 | 188 | 20 | 12 | 341
  Non-Hispanic African American | 0 | 0 | 8 | 1 | 3 | 12
  Non-Hispanic Asian | 1 | 1 | 0 | 1 | 0 | 3
  Hispanic, White | 0 | 0 | 3 | 0 | 0 | 3
  Non-Hispanic Native Am | 1 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 55 | 69 | 199 | 23 | 15 | 361
Disease [Count of Participants; unit: Participants]
  Acute myeloid leukemia | 17 | 25 | 89 | 13 | 3 | 147
  Acute lymphoblastic leukemia | 2 | 30 | 16 | 5 | 1 | 54
  Chronic myeloid or lymphocytic leukemia | 14 | 7 | 14 | 0 | 2 | 37
  Hodgkin or Non-Hodgkin lymphoma or multiple myeloma | 6 | 2 | 56 | 4 | 4 | 72
  Myelodysplastic syndrome or myeloproliferative disorder | 15 | 3 | 23 | 1 | 1 | 43
  Severe Aplastic anemia | 1 | 2 | 1 | 0 | 3 | 7
  Solid Tumor | 0 | 0 | 0 | 0 | 1 | 1
Risk group [Count of Participants; unit: Participants]
  Standard | 32 | 42 | 73 | 10 | 4 | 161
  High | 23 | 27 | 126 | 13 | 11 | 200

OUTCOME MEASURES:

1. Primary Outcome: CR Rate
Description: Rate of Complete Remission by Day +100
Time Frame: day 100
Measure: Count of Participants; unit: Participants
Arm/Group | BuCy | CyTBI | FluMel | VpCyTBI | Other
Number analyzed (Participants) | 55 | 69 | 199 | 23 | 15
Participants | 42 | 55 | 134 | 18 | 7

2. Secondary Outcome: Toxicity/TRM at Day 100
Description: Death due to treatment related causes before day +100 after BMT
Time Frame: Day +100
Measure: Count of Participants; unit: Participants
Arm/Group | BuCy | CyTBI | FluMel | VpCyTBI | Other
Number analyzed (Participants) | 55 | 69 | 199 | 23 | 15
Participants | 3 | 4 | 31 | 4 | 4

3. Secondary Outcome: 4 Year PFS
Description: progression free survival estimate at 4 years post BMT (events are disease progression/relapse and death due to any cause)
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BuCy | CyTBI | FluMel | VpCyTBI | Other
Number analyzed (Participants) | 55 | 69 | 199 | 23 | 15
percentage of participants | 49.1 [36 to 62.2] | 52.2 [40.4 to 64] | 33.2 [26.7 to 39.7] | 26.1 [8.1 to 44.1] | 40 [15.3 to 64.7]

4. Secondary Outcome: 4 yr OS
Description: Overall survival estimate at 4 years post BMT
Time Frame: 4-year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BuCy | CyTBI | FluMel | VpCyTBI | Other
Number analyzed (Participants) | 55 | 69 | 199 | 23 | 15
percentage of participants | 56.4 [43.3 to 69.5] | 56.5 [44.7 to 68.3] | 38.2 [31.5 to 44.9] | 39.1 [19.1 to 59.1] | 53.3 [28 to 78.6]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | BuCy | CyTBI | FluMel | VpCyTBI | Other
All-Cause Mortality (participants affected / at risk) | 30/55 | 36/69 | 150/199 | 19/23 | 9/15
Serious Adverse Events (participants affected / at risk) | 11/55 | 10/69 | 62/199 | 6/23 | 4/15
Other Adverse Events (participants affected / at risk) | 25/55 | 35/69 | 100/199 | 6/23 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BuCy (N=55) | CyTBI (N=69) | FluMel (N=199) | VpCyTBI (N=23) | Other (N=15)
1 yr TRM (Investigations) | 11 (11) | 10 (10) | 62 (62) | 6 (6) | 4 (4) — death due to transplant related causes before 1 year after BMT
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BuCy (N=55) | CyTBI (N=69) | FluMel (N=199) | VpCyTBI (N=23) | Other (N=15)
acute graft-versus-host disease (Blood and lymphatic system disorders) | 25 (25) | 35 (35) | 100 (100) | 6 (6) | 9 (9) — overall grade II to IV acute graft versus host disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT00003816/Prot_SAP_000.pdf